CLINICAL TRIAL: NCT06226532
Title: Effect of Lidocaine Sprayed at the Laryngeal Inlet and Endotracheal Tube Cuff Versus Intravenous Lidocaine for Attenuating Hemodynamic Response During Laryngoscopy and Intubation in Neurosurgical Patients
Brief Title: Effect of Lidocaine Sprayed for Attenuating Hemodynamic Response During Laryngoscopy and Intubation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Nattawadee Phokaw, MD, Principal investigator, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE661362
Record Dates: First submitted 2024-01-02; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Laryngoscopy; Intubation; Hemodynamics; Neurosurgery; Lidocaine
Keywords: Lidocaine; Laryngoscopy and intubation; Hemodynamics; Neurosurgery

STUDY DESIGN:
Intervention Model Description: 1. Group SL: 10%lidocaine spray total 8 puffs at laryngoscopes blade and endotracheal tube cuff.
  2. Group IL: 2% lidocaine intravenous 1.5 mg/kg, not exceed 80 mg equally to spray group.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group SL (Experimental): 10%lidocaine spray total 8 puffs at laryngoscopes blade and endotracheal tube cuff, 4 puffs each.
  Interventions: Drug: lidocaine spray
- Group IL (Active Comparator): 2% lidocaine intravenous 1.5 mg/kg, not exceed 80 mg equally to spray group.
  Interventions: Drug: Intravenous Lidocaine

INTERVENTIONS:
Drug: lidocaine spray — Group SL: Spray 10% lidocaine for 4 puffs at the endotracheal tube cuff, also prepare for spray at the laryngeal inlet for 4 puffs (total approximately 1.5mg/kg)
  Other Names: 10% lidocaine spray
  Arms: Group SL
Drug: Intravenous Lidocaine — 2% lidocaine 1.5 mg/kg IV will be given 2 minutes after cisatracurium injection (3 minutes prior intubation).
  Other Names: 2%Intravenous Lidocaine
  Arms: Group IL

SUMMARY:
The goal of this clinical trial is to to evaluate the efficacy of lidocaine sprayed at the laryngeal inlet combined with the endotracheal tube cuff compare with intravenous lidocaine on the hemodynamic response to laryngoscopy and intubation in patients undergoing elective neurological procedures during general anesthesia with total intravenous technique.

The main question it aims to answer is:

- Does topical lidocaine sprayed at the laryngeal inlet combined with the endotracheal tube cuff have more effect on stabilizing hemodynamic responses to laryngoscopy and intubation than intravenous lidocaine, in neurosurgical patients who undergo general anesthesia with total intravenous technique?

Participants will be recruited and randomized to receive either lidocaine spray (Group SL) or intravenous lidocaine (group IL) to blunt hemodynamic response to laryngoscopy and intubation.

DETAILED DESCRIPTION:
Anesthetic protocol

* Preoperative

  * After the informed consent, all eligible patients will be fasting after midnight as it is an elective procedure.
  * No preoperative sedatives or analgesics were administered.
* Intraoperative Pre-induction phase

  * Standard monitors of electrocardiogram, noninvasive blood pressure (NIBP) is measured at upper extremity with BP cuff bladder length ≥ 80% and width ≥40% of patient's arm circumference and pulse oximeter were attached.
  * BIS (Bispectral index) was monitored
  * Hemodynamic baseline values of heart rate (HR), systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean arterial pressure (MAP) were recorded before the induction.

Intervention: prepared before induction anesthesia.

* Group SL: Spray 10% lidocaine for 4 puffs at the endotracheal tube cuff, also prepare for spray at the laryngeal inlet for 4 puffs (total approximately 1.5mg/kg).
* Group IL: 2% lidocaine 1.5 mg/kg IV will be given 2 minutes after cisatracurium injection (3 minutes prior intubation).

Induction phase

* Preoxygenation 100% oxygen, flow 6 liters per minute, for 3-5 minutes, target end tidal oxygen more than 90%
* Medication before the induction of anesthesia includes fentanyl 1.5 mcg/kg IV.
* General anesthesia will be induced with propofol target-controlled infusion (TCI) 4-6 mcg/ml IV, followed by cisatracurium 0.15 mg/kg IV for intubation.
* Bag mask ventilation will be started.
* The arterial line will be canulated before direct laryngoscopy and intubation and arterial line pressure transducer will be levelled at the phlebostatic axis and calibrate with NIBP.
* Intervention: Group IL: 2% lidocaine 1.5 mg/kg IV was given 2 minutes after cisatracurium injection.
* Direct laryngoscopy and tracheal intubation were done by an anesthesiologist, 1st (6 months experience), 2nd, and 3rd years anesthesiology resident.

At 5 minutes after cisatracurium injection, direct laryngoscopy will be performed, and spray 10%lidocaine directly to the epiglottis for 4 puffs for SL group.

* Tracheal intubation will be performed.
* The bispectral index (BIS) target range during intubation is 40 to 60.
* The hemodynamic parameters including mean arterial pressure(MAP) in mmHg, systolic blood pressure(SBP) in mmHg, diastolic blood pressure(DBP) in mmHg and heart rate(HR) in beats per minutes(bpm) and BIS will record during the peri-intubation period

All the adverse events (cough, pulmonary aspiration, desaturation, hypotension, hypertension, tachycardia, bradycardia, and arrythmia) will be noted as yes or no.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old
2. American Society of Anesthesiologists (ASA) physical status classification I-II

Exclusion Criteria:

1. History of lidocaine allergy
2. Predicted difficult airways
3. Body mass index > 35 kilograms per meter squared
4. Risk aspiration
5. Baseline hemodynamic instability; heart rate < 50 bpm, heart rate > 120 bpm, blood pressure < 90/60 mmHg, blood pressure > 160/90 mmHg
6. Underlying disease: epilepsy, cardiovascular disease, heart failure, impaired cardiac function, severe renal dysfunction, impaired hepatic function, peripheral vascular disease
7. Pregnancy
8. Cerebral aneurysm, Arteriovenous malformation, Tumor size > 4 centimeters, Brain herniation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Changing in mean arterial pressure (MAP) during the peri-intubation period | T0: Baseline at operating room, T1: immediately after cisatracurium injection, T2: During direct laryngoscopy, T3: During intubation, T4-T9: repeated measurement every 1 minute until 6 minute after intubation
  Mean arterial pressure was recorded in mmHg by the anesthesiologist
Changing in blood pressure (BP) during the peri-intubation period | T0: Baseline at operating room, T1: immediately after cisatracurium injection, T2: During direct laryngoscopy, T3: During intubation, T4-T9: repeated measurement every 1 minute until 6 minute after intubation
  Blood pressure was recorded in mmHg by the anesthesiologist
Changing in heart rate (HR) during the peri-intubation period | T0: Baseline at operating room, T1: immediately after cisatracurium injection, T2: During direct laryngoscopy, T3: During intubation, T4-T9: repeated measurement every 1 minute until 6 minute after intubation
  Heart rate was recorded in bpm by the anesthesiologist

SECONDARY OUTCOMES:
Incidence of adverse event during laryngoscopy and intubation procedure | During laryngoscopy and intubation procedure
  Adverse events were recorded by the anesthesiologist. The adverse events included coughing, desaturation, aspiration, hypotension, hypertension, tachycardia, and bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Nattawadee Phokaw, MD, Principal Investigator — Department of anesthesiologist, Faculty of Medicine, Khon Kaen University
Locations (1):
- Khon Kaen University, Nai Muang, KhonKaen, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Researcher who required more information for further study

REFERENCES:
- [Background] Ismail SA, Bisher NA, Kandil HW, Mowafi HA, Atawia HA. Intraocular pressure and haemodynamic responses to insertion of the i-gel, laryngeal mask airway or endotracheal tube. Eur J Anaesthesiol. 2011 Jun;28(6):443-8. doi: 10.1097/EJA.0b013e328345a413. PMID 21455075
- [Background] Basali A, Mascha EJ, Kalfas I, Schubert A. Relation between perioperative hypertension and intracranial hemorrhage after craniotomy. Anesthesiology. 2000 Jul;93(1):48-54. doi: 10.1097/00000542-200007000-00012. PMID 10861145
- [Background] Tada Y, Wada K, Shimada K, Makino H, Liang EI, Murakami S, Kudo M, Kitazato KT, Nagahiro S, Hashimoto T. Roles of hypertension in the rupture of intracranial aneurysms. Stroke. 2014 Feb;45(2):579-86. doi: 10.1161/STROKEAHA.113.003072. Epub 2013 Dec 26. PMID 24370755
- [Background] Khan FA, Ullah H. Pharmacological agents for preventing morbidity associated with the haemodynamic response to tracheal intubation. Cochrane Database Syst Rev. 2013 Jul 3;2013(7):CD004087. doi: 10.1002/14651858.CD004087.pub2. PMID 23824697
- [Background] Gerlach AT, Murphy CV. Dexmedetomidine-associated bradycardia progressing to pulseless electrical activity: case report and review of the literature. Pharmacotherapy. 2009 Dec;29(12):1492. doi: 10.1592/phco.29.12.1492. PMID 19947809
- [Background] Tam S, Chung F, Campbell M. Intravenous lidocaine: optimal time of injection before tracheal intubation. Anesth Analg. 1987 Oct;66(10):1036-8. No abstract available. PMID 3631567
- [Background] Shribman AJ, Smith G, Achola KJ. Cardiovascular and catecholamine responses to laryngoscopy with and without tracheal intubation. Br J Anaesth. 1987 Mar;59(3):295-9. doi: 10.1093/bja/59.3.295. PMID 3828177
- [Background] Lee SY, Min JJ, Kim HJ, Hong DM, Kim HJ, Park HP. Hemodynamic effects of topical lidocaine on the laryngoscope blade and trachea during endotracheal intubation: a prospective, double-blind, randomized study. J Anesth. 2014 Oct;28(5):668-75. doi: 10.1007/s00540-014-1812-z. Epub 2014 Mar 12. PMID 24619576